CLINICAL TRIAL: NCT07263685
Title: Retrospective Chart Review Study Evaluating Clinical Effectiveness and Impact on Quality of Life Among Patients Who Initiated Long-term Prophylaxis With Takhzyro® in a Real-World Setting in the Kingdom of Saudi Arabia - the REFLEQT-KSA Study (Retrospective Evaluation Focusing on Lanadelumab's Effectiveness and Impact on Quality of Life in The Kingdom of Saudi Arabia)
Brief Title: A Study of Lanadelumab in Teenagers and Adults With Hereditary Angioedema (HAE) in the Kingdom of Saudi Arabia
Status: Not yet recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-743-4037
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: Drug Therapy
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with HAE-C1INH-Type 1 or HAE-C1INH-Type 2: All participants diagnosed with HAE-C1INH type 1 or type 2 will be included, and retrospective clinical data will be collected from patient medical records between 01 September 2025 and 28 February 2026. Participants who received Takhzyro® during the eligibility period beginning in 2021 will be observed across two periods: a pre-index period, defined as the time before the first dose of Takhzyro® (index date), used to establish baseline characteristics and disease activity, and a post-index period, defined as at least 6 months following the index date, used to assess treatment outcomes. The index date is defined as the date of the first Takhzyro® administration during the eligibility period.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a non-interventional study.

SUMMARY:
Hereditary angioedema (HAE) is a rare condition. It causes sudden swelling under the skin and inside the body, like in the belly, throat, or genitals. This swelling happens because of a temporary leak in blood vessels but does not cause itching or hives. HAE is classified based on the amount of a protein in the blood called C1 inhibitor (C1INH): HAE with normal C1INH levels (HAE-nC1INH) and HAE with limited or insufficient C1INH levels (HAE-C1INH); HAE-C1INH can be divided into Type 1, with low levels of C1INH, and Type 2, in which the protein is there, but does not work properly. This study will concentrate on people with HAE-C1INH Type 1 or 2 who have received Takhzyro® (lanadelumab) as prophylactic treatment for at least half a year (6 months). Prophylactic means that treatment is given to prevent the happening of HAE attacks.

The main goal of the study is to see how well Takhzyro® works in everyday life to reduce the condition's activity after 6 months of treatment, or 12 months (if data is available). This will be measured by checking the change of the HAE activity from before treatment to after 6 months of treatment.

The study design will permit a study follow-up of up to 12 months following the index event (i.e. date of first dose administration of Takhzyro®) unless the patient discontinues the index treatment, dies or is lost to follow-up within this timeframe. Chart abstractions will only occur once patients have at least 6 months' duration between the index event date and the date of chart abstraction initiation. Other goals are to find out how a person's quality of life changes after using Takhzyro® for 6 months, how often they had attacks before and after treatment and to learn which factors may have an impact on the treatment.

The study will only look at data already existing in the participants' medical records. No treatment will be given as part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is diagnosed with HAE-C1INH-Type 1 or HAE-C1INH-Type 2 and initiated on long-term prophylaxis (LTP) with Takhzyro® (lanadelumab).
2. Participant is aged greater than or equal to (>=) 12 years at the time of Takhzyro® initiation.
3. Participant has received at least 6 months of continuous treatment with Takhzyro® before data abstraction.

Exclusion Criteria:

1. Participants who have normal C1INH function or HAE-nC1INH (formerly type III HAE).
2. Participants who discontinued Takhzyro® before completing 6 months of treatment.
3. Participants with insufficient or incomplete medical records which prevent the assessment of baseline HAE-AS at the time of Takhzyro® initiation, as well as 6 months HAE-AS after treatment initiation.
4. Participants who are participating in an interventional clinical trial involving other HAE-C1INH treatments during the observation period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents and adult participants with HAE-C1INH-Type 1 or HAE-C1INH-Type 2 treated with lanadelumab in routine clinical setting in the Kingdom of Saudi Arabia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in HAE- Activity Score (AS) From Pre to Post Index Period | Up to 6 Months
  HAE-AS is a patient-reported outcome (PRO) instrument used to measure the activity of HAE. It comprises 12 items assessing factors like attack frequency, emergency visits, and impact on daily life over a recall period. A higher HAE-AS score indicates greater disease activity. A score of 13 or higher suggests severe HAE activity, while a score below 12 indicates mild or low activity.

SECONDARY OUTCOMES:
Change in Quality of Life (QoL) Scores From Pre to Post Index Period | Up to 6 months
  A study-specific quality-of-life (QoL) score will be developed. This custom score will be derived from select parameters conceptually aligned with the domains of the validated Angioedema (AE)-QoL (functioning, fatigue/mood, fear/shame, and nutrition), as captured in the available participant records. The goal is to approximate core aspects of health-related quality of life relevant to participants with recurrent angioedema, while ensuring feasibility and compliance within the constraints of retrospective data collection.
Change in HAE-C1INH Attack Frequency (number/month) From Pre to Post Index Period | Up to 6 months
  HAE attack is defined as a discrete episode during which the participant progresses from no angioedema to symptoms of angioedema. A "change in HAE-C1INH attack frequency" refers to the reduction in the number of HAE attacks (number per month) after the implementation of treatments.
Number of Participants Categorized by Demographic and Clinical Predictors of Treatment Response | From Baseline up to end of study (up to 6 months)
  Number of participants will be reported by baseline demographic (age, sex) and clinical characteristics (disease duration, baseline attack frequency). The relationship between these characteristics and change from baseline in HAE-AS score and attack frequency will be further explored using regression analysis, provided sufficient sample size and model stability.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/ba5551a2b34748ad??page=1&idFilter=TAK-743-4037